CLINICAL TRIAL: NCT05158218
Title: Robotic Exoskeleton Gait Training in Adolescents With Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Father Flanagan's Boys' Home (Other)
Responsible Party: Principal Investigator, Max Kurz, Director of PoWER Lab, Father Flanagan's Boys' Home
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-12-XP
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Gait Therapy; Mobility; Robotic Exoskeleton
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Cerebral Palsy participants will undergo baseline mobility/brain imaging/cognitive testing, receive traditional gait therapy, and then repeat mobility/brain imaging testing.
  Cerebral Palsy participants will undergo baseline mobility/brain imaging/cognitive testing, receive gait therapy utilizing robotic exoskeleton, and then repeat mobility/brain imaging testing.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebral Palsy Youth/Young Adults Physical Therapy (Active Comparator): Baseline and 8 week assessments; 8 week gait therapy
  Interventions: Behavioral: Physical Therapy
- Cerebral Palsy Youth/Young Adults Robotic Exoskeleton (Experimental): Baseline and 8 week assessments; 8 week gait therapy using robotic exoskeleton
  Interventions: Behavioral: Robotic Exoskeleton Gait Therapy

INTERVENTIONS:
Behavioral: Robotic Exoskeleton Gait Therapy — The training protocol will consist of 24-treatment sessions that will be performed 3 times-a-week for an 8-week period. All therapeutic exercises will be performed under the direction of a licensed physical therapist. Any sessions missed will be added on to the 8-week period. Each intervention session will be completed in a 60-minute sessions with rests as needed. The key components of the therapy will include: 1) optimally challenging activities of variable intensity that emphasize motor planning and problem solving that requires altering the leg kinematics to meet the environmental and task constraints, 2) task specific overground movements that promote building a repertoire of mobility strategies that can be utilized in the community, and 3) motor tasks requiring active control that increase participant therapeutic engagement. An overhead body weight support system or a gait-belt may be used for some individuals during the robotic exoskeleton gait training blocks.
  Arms: Cerebral Palsy Youth/Young Adults Robotic Exoskeleton
Behavioral: Physical Therapy — The training protocol will consist of 24-treatment sessions that will be performed 3 times-a-week for an 8-week period. All therapeutic exercises will be performed under the direction of a licensed pediatric physical therapist. Any sessions missed will be added on to the 8-week period. Each intervention session will consist of over-ground gait activities that will be completed in a 60 minute session with rests as needed. The key ingredients of the therapy will include: 1) activities of adequate intensity that promote gait adaptation and gait speed sustainment, 2) exploratory activities that enhance the somatosensory experience through rich/novel movement, and 3) optimally challenging activities that emphasize planning and problem solving that requires altering the leg kinematics to meet the environmental and task constraints. An overhead body weight support system or a gait-belt may be used for some individuals during the gait training blocks
  Arms: Cerebral Palsy Youth/Young Adults Physical Therapy

SUMMARY:
The study design will consist of a cohort of adolescents and young adults with cerebral palsy (CP) that will undergo a gait training protocol. All participants will complete MEG baseline brain imaging measures of their sensorimotor cortical activity, MRI brain/spinal cord imaging (previous MRI or template brain may be substituted), neurophysiological tests of the spinal cord H-reflex, and a series of mobility clinical tests.

After completing the baseline tests, the participants with CP will undergo the therapeutic gait training using either traditional physical therapy or utilizing a robotic exoskeleton. After completing all of the therapeutic gait training sessions, the participants will repeat the same assessments that were completed at baseline. The two groups will be compared based on the assessments for therapeutic outcomes.

DETAILED DESCRIPTION:
Cerebral palsy (CP) results from a perinatal brain injury and is one of the most prevalent and costly pediatric neurologic conditions in the United States that often results in mobility deficits. The investigator's extensive experimental work has been focused on developing a therapeutic gait training protocol that will improve the long-term mobility of adolescents and young adults with CP. Robotic exoskeletons have gained recent attention in the therapeutic community as a high-tech option for assisting with over-ground mobility of various patient populations. The goal of this investigation is to take a fresh new approach on how robotic exoskeletons can be used in a therapeutic setting. As opposed to using them as a compensation tool, we are proposing to use them to perturb the legs to drive beneficial neuroplasticity in the key brain areas that govern the leg motor actions. Essentially, we predict that the neuroplastic changes promoted by the exoskeleton gait training protocol will lead to more robust clinical outcomes than what is seen by gait training alone. The aims of this study will: (1) determine if individuals with CP that undergo a robotic exoskeleton gait training protocol have larger mobility improvements compared to those that undergo gait training alone, (2) determine if individuals that undergo a robotic exoskeleton gait training protocol have larger improvements in key brain areas involved in motor planning and execution of the leg motor actions compared to those that undergo gait training alone, and (3) determine if individuals with CP that undergo a robotic exoskeleton gait training protocol have larger mobility improvements compared to those that undergo gait training alone. It is hypothesized after exoskeleton gait training participants will demonstrate substantially greater improvements in their 10-meter walk speed, one-minute walk test, and Functional Gait Assessment scores. Additionally, following exoskeleton training, the sensorimotor cortical activity will be significantly different from what is seen in those receiving gait training alone. Furthermore, the degree of brain activity changes will be related to the extent of the mobility improvements seen after completing the exoskeleton gait training protocol. Briefly, the study design consists of a cohort of adolescents and young adults with CP that will initially undergo MEG brain imaging, MRI spinal cord imaging, neurophysiological tests of the spinal cord interneuronal circuitry, and clinical mobility assessments. After completing the baseline tests, the participants will undergo either traditional therapeutic gait training or utilize the robotic exoskeleton gait therapy. Upon completion of the treatment program, participants will undergo the same baseline assessments. The results from the post therapy outcomes will be compared between the two groups: traditional gait therapy and robotic exoskeleton.

ELIGIBILITY:
Inclusion Criteria:

* For Cerebral Palsy participants:

  * Cerebral Palsy diagnosis
* For Non-Cerebral Palsy Controls:

  * No known atypical neurodevelopment (e.g autism, Down Syndrome, ADHD, etc.)

Exclusion Criteria:

* No orthopedic surgery in the last 6 months or metal in their body that would preclude the use of an MRI.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mobility Test Time | Baseline (CP and Neurotypical) and 8 weeks (CP)
  The participant will be asked to perform a series of timed (in seconds) 10-meter walking tasks.
Change in Time for Community Ambulation | Baseline (CP and Neurotypical) and 8 weeks (CP)
  The participants will walk along a 400 meter course laid out on the Boys Town campus that incorporates uphill/downhill grades, stairs, curbs, grass and uneven surfaces. The time (in seconds) to complete the course will be used as an outcome variable.
Change in Time for "Timed Up and Go" | Baseline (CP and Neurotypical) and 8 weeks (CP)
  The participant will start the test by sitting on a bench. The time (in seconds) it takes the participant to stand-up, walk to a line on the floor that is 3-meters away and return back to sitting on the bench will be the outcome measure.
Change in Selective Control Assessment of the Lower Extremity | Baseline (CP and Neurotypical) and 8 weeks (CP)
  This is a clinical assessment where the participant is asked to isolate and move the lower extremity joints. The examiner grades the amount of movement and the ability of the participant to isolate the control. A grade of 0 indicates the participant cannot move the joint, 1 indicates the participant can move the joint but it is impaired, and 2 indicates normal movement of the joint.
Change in Level of Spasticity | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Modified Ashworth: This is a clinical assessment where the therapist passively moves the participant's joints and rates the level of spasticity. Scores range from 0-5, where 0 indicates no tone, 5 indicates rigidity.
Change in Isolation of Movement | Baseline (CP and Neurotypical) and 8 weeks (CP)
  This is a clinical assessment where the participant is asked to isolate and move the lower extremity joints. The examiner grades the amount of movement and the ability of the participant to isolate the control. A grade of 0 indicates the participant cannot move the joint, 1 indicates the participant can move the joint but it is impaired, and 2 indicates normal movement of the joint.
Change in Brain Activity in Sensory Cortices | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Magnetoencephalogram (MEG) or electroencephalogram (EEG) scan: The frequency bands of interest include theta (4-8 Hz), alpha (8-12 Hz), beta(15-30 Hz) and gamma (>30 Hz).
Change in Motor Response | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Percutaneous electrical stimulations of the femoral nerve applied via an anode that is positioned on the patella and a cathode that is positioned on the popliteal fossa will be applied to the right leg. A wireless surface EMG sensor positioned on the soleus will measure the motor response. The muscular (M-wave) will be assessed while resting and walking.
Change in Hoffmann Reflex | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Percutaneous electrical stimulations of the femoral nerve applied via an anode that is positioned on the patella and a cathode that is positioned on the popliteal fossa will be applied to the right leg. A wireless surface EMG sensor positioned on the soleus will measure the Hoffmann reflex. The spinal reflexes (H-wave) will be assessed while resting and walking.

SECONDARY OUTCOMES:
Cognitive related changes induced via physical therapy -Wide Range Assessment of Memory and Learning (WRAML) | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Subtests: Finger Windows, Picture Memory, Symbolic Working Memory:
Cognitive related changes induced via physical therapy - D2 - Test of Attention | Baseline (CP and Neurotypical) and 8 weeks (CP)
  A neuropsychological measure of selective and sustained attention in addition to visual scanning speed. Participants are tasked with crossing out any letter "d" with two marks around above it or below it in any order, in a mix of other letters and with various numbers of marks around them. Viable for young children and adults.
Cognitive related changes induced via physical therapy - Trail Making A+B | Baseline (CP and Neurotypical) and 8 weeks (CP)
  A neuropsychological test of visual attention and task switching. The subject is tasked to connect a set of numbered 25 dots as quickly as possible while still maintaining accuracy, with the second test increasing in cognitive load by introducing letters as well. Viable for young children and adults.
Cognitive related changes induced via physical therapy - WAIS-IV Digit Span - Youth + Adult | Baseline (CP and Neurotypical) and 8 weeks (CP)
  A subtest of the Wechsler Memory Scales (WMS), subjects are read a sequence of numbers and asked to repeat the same sequence back to the examiner in order (forward span) or in reverse order (backward span) to measure short term memory capacity in young children and adults.
Cognitive related changes induced via physical therapy - Stroop Test - Youth + Adult | Baseline (CP and Neurotypical) and 8 weeks (CP)
  A neuropsychological test that assesses the ability to inhibit cognitive interference during the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute (the Stroop Effect). The Stroop Effect is the delay in reaction time between congruent and incongruent stimuli, Such that a mismatch between the name of a color (e.g., "blue", "green", or "red") and the color it is printed on (i.e., the word "red" printed in blue ink instead of red ink).
Cognitive related changes induced via physical therapy - Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) Questionnaire | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Children with severe developmental disabilities are often dependent on parents/caregivers for much of their daily needs. These children often have multiple co-morbid conditions which can have a significant impact on their overall health and quality of life. Interventions are aimed at preserving or improving their health, comfort and quality of life and to facilitate caregiving. CP CHILD is an instrument that aims to measure these phenomena. Respondents rate a number of areas including the difficulty of activities for their child (Scale ranging from 0-Not Possible to 6-No problem at all) and choose the level of assistance needed to perform these activities (Scale ranging from 0-Total to 3-Independent), how often their child experience pain or discomfort (Scale ranging from 0-Every day to 5-None of the time) and intensity (0-Severe to 3-None), importance of items in child's quality of life (0-Least Important to 5-Most Important), and overall health of child (0-Very Poor to 5-Excellent).
Cognitive related changes induced via physical therapy - Silver Linings Questionnaire - Adapted for CP | Baseline (CP and Neurotypical) and 8 weeks (CP)
  A survey measure that examines the extent to which people believe their illness - in this case the questionnaire has been adapted to individuals with CP, has had a positive benefit despite the negative consequences of having CP. Participants indicate the extent to which they agree or disagree with each statement by circling a number between 5 "strongly agree" and 1 "strongly
Cognitive related changes induced via physical therapy - Child and Adolescent Sleep Checklist (CASC) | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Tool designed to identify sleep habits and to make a screening of sleep problems among preschoolers, elementary school children, and high school students.
Cognitive related changes induced via physical therapy - PEDS QL Fatigue Questionnaire (Acute) | Baseline (CP and Neurotypical) and 8 weeks (CP)
  The PedsQL Multidimensional Fatigue Scale is a symptom-specific instrument to measure fatigue across pediatric populations. It measures cognitive fatigue which focuses on problems with memory and attention, areas known to be affected in children with CP, on a scale ranging from 0-if it is never a problem and 4-if it is almost always a problem.
Cognitive related changes induced via physical therapy - Pittsburgh Sleep Quality Index (PSQI) | Baseline (CP and Neurotypical) and 8 weeks (CP)
  An effective instrument used to measure the quality and patterns of sleep in adults.
Cognitive related changes induced via physical therapy - MacArthur Scale of Subjective Social Status Youth + Adult | Baseline (CP and Neurotypical) and 8 weeks (CP)
  Adult Version: This tool for adults, uses a pictorial representation of a symbolic ladder, developed to capture the common sense of social status based on usual socioeconomic status indicators. It has the additional advantage to allow comparisons between studies conducted in different populations.

CONTACTS AND LOCATIONS:
Overall Officials: Max J Kurz, PhD, Principal Investigator — Father Flanagan's Boys' Home
Locations (1):
- Boys Town National Research Hospital, Boys Town, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI and all of the investigators have made a commitment to publish, in a timely manner, all of the relevant scientific information that they will derive during this project. Deidentified data will be made available upon reasonable request to the Principal Investigator (Dr. Kurz).
Supporting Information: Study Protocol, CSR
Time Frame: Upon completion of study and data analysis.
Access Criteria: Contact Dr. Kurz